CLINICAL TRIAL: NCT06044701
Title: The Effect of Hologram Fan and Bubble Machine Use on Pain and Fear During Intravenous Blood Collection in Children
Brief Title: Pain and Fear During Intravenous Blood Collection in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, CANSU OZTURK, Principal investigator, Ege University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: EU-SBE-CO-01
Record Dates: First submitted 2023-05-05; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Procedural Pain
Keywords: fear; pain; pediatrics; hologram; bubble-blowing; invasive procedures
MeSH Terms: conditions — Pain, Procedural; Pain

STUDY DESIGN:
Intervention Model Description: The randomization method:
  Children who meet the sample selection criteria will be randomly assigned to three groups: bubble machine group (n=55), hologram fan group (n=55) and control group (n=55). The assignment of individuals to the study groups will be carried out by block randomization method and the blocks will be formed according to age groups (3-7 years / 8-12 years: 2 blocks). The confidentiality of assigning to groups will be ensured by a table of numbers created on the computer by a person independent of the research.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hologram fan (Active Comparator): Hologram fan application during blood collection process
  Interventions: Other: Hologram Distraction Technique
- Bubble machine (Active Comparator): Bubble machine application during blood collection
  Interventions: Other: Bubble Machine Distraction Technique
- Control Group (No Intervention): Performing routine application during the blood collection process

INTERVENTIONS:
Other: Hologram Distraction Technique — Hologram fan application during blood collection process
  Other Names: Hologram Fan
  Arms: Hologram fan
Other: Bubble Machine Distraction Technique — Bubble machine application during blood collection
  Other Names: Bubble machine
  Arms: Bubble machine

SUMMARY:
Medical procedures can cause significant stress and anxiety for children and parents, impacting their overall hospital experience. Numerous studies have demonstrated that techniques aimed at diverting attention during procedures can effectively reduce pain and fear. Considering the rapid advancements in technology and the strong connection between Generation Z children and technology, this study aims to explore the use of hologram technology through a hologram fan and the traditional method of bubble blowing as interventions to assess their impact on pain and fear levels during intravenous blood collection in children.

The study design will follow a randomized controlled trial approach. The sample will consist of patients between the ages of 3 and 12 who meet the sampling criteria and receive outpatient care at the pediatric stem cell outpatient treatment unit between April 2022 and February 2024. Data will be collected using a researcher-prepared form containing introductory information and child pain, fear, and emotional indicator scales for which appropriate permissions have been obtained. The blood collection process will be performed by the unit's nurse, and the observer nurse will complete the scales.

Descriptive statistics, such as mean, standard deviation (median, minimum, maximum), frequency, and percentage values, will be used for data analysis. IBM SPSS Statistics 25.0 (IBM SPSS Statistics for Windows, Version 25.0. Armonk, NY: IBM Corp.) will be employed for data analysis. A significance level of 0.05 will be used for all statistical analyses.

Regenerate response Keywords: Fear, pain, pediatrics, hologram, bubble-blowing, invasive procedures

DETAILED DESCRIPTION:
Pediatric clinics often subject infants and children to painful medical procedures. These interventions include blood collection, intramuscular and intravenous injections, which can induce pain and fear in children. The experience of pain during medical procedures has long-term effects and can shape a person's approach to healthcare in the future. While evidence-based practices exist to address interventional pain in the pediatric population, they may not always be sufficient in practice. As technology advances, there is growing interest in innovative methods to reduce pain, alongside commercially available products.

Distraction techniques have been proven effective in reducing acute pain in children during needle interventions. Distraction aims to redirect the child's attention to another stimulus, based on the understanding that the brain has limited capacity to focus on pain. Nurses and healthcare workers play a crucial role in alleviating children's fear of medical procedures, as they are often the first point of contact and provide ongoing care.

In addition to traditional methods such as watching cartoons, inflating balloons, and playing music, innovative techniques have emerged. One such method is the use of bubble machines, which produce bubbles using blowing and spraying systems. Studies have shown that bubble blowing can effectively reduce pain intensity during phlebotomy in children aged 3-6 years. Other studies have recommended using bubble blowing alongside devices like Buzzy to reduce pain severity during phlebotomy and intramuscular injections.

Considering the current pandemic situation, the use of bubble machines has gained attention as a potentially more effective distraction method than balloon blowing, as it reduces the risk of infection and provides a greater number of bubbles in the environment. Moreover, hologram technology has gained popularity in our daily lives. Holography refers to three-dimensional projections that can be seen without special equipment. It has the potential to revolutionize medicine by providing realistic and immersive experiences. However, there is a lack of studies exploring the application of hologram technology in reducing pain during medical procedures, particularly in the nursing literature. It is believed that this technology can effectively distract children during painful interventions.

Technological advancements, including hologram technology, have the potential to significantly impact the healthcare sector. By utilizing such applications, especially for diversion and comfort in pediatric pain management, healthcare professionals can improve the overall experience of children. The use of technology can also enhance efficiency and service quality in healthcare, benefiting patients of all age groups.

In this context, the present study aims to investigate the use of hologram fans and bubble machines to divert attention, reduce fear and pain levels, and improve compliance during intravenous blood collection in children. This unique study, which incorporates hologram technology, aims to contribute to the existing literature. Similar to bubble machines, bubble blowing toys have been studied and have shown attention-grabbing effects. Therefore, this study is necessary to explore the effects of hologram fans and bubble machines on children's pain and fear levels during intravenous blood collection, a highly stressful procedure for both children and parents, and to introduce new methods to the literature on this topic.

Hologram: The word hologram means "three-dimensional image recording system" in Turkish. Hologram is the name given to the picture obtained by the use of coherent laser beams. Along with the intensity of light, the hologram allows an object to be seen in three dimensions by recording the direction of the light waves.

Hologram Fan: A hologram fan is one of the industrial electronic products that creates an illusion of 3D objects circling in the air. The fan rotates too fast to be seen with the naked eye, resulting in a transparent background for the projected object.

Bubble Machine: These are the systems used in blowing sequencing by adding liquid mixtures specially prepared for bubbles to the machine chamber. Warm-up times are provided in 5-10 seconds, the machines provide use on blowing and spraying systems and the production of bubbles and their release to the space used.

Purpose of the Study: The aim of this study was to investigate the effect of hologram fan and bubble machine use on pain and fear levels during blood collection process in children who applied to Pediatric Stem Cell Transplantation Polyclinic at Ege University Children's Hospital.

Hypotheses H1: The use of a hologram fan reduces interventional pain during the blood collection process.

H2: The use of a bubble machine reduces interventional pain during the blood collection process.

H3: The use of a hologram fan reduces the fear of interference during the blood collection process.

H4: The use of a bubble machine reduces the fear of interference during the blood collection process.

H5: The use of a hologram fan affects the emotional behavior scale score during the blood collection process.

H6: The use of a bubble machine affects the emotional behavior scale score during the blood collection process.

Wong- Baker Faces Pain Scale The scale consists of six black and white faces, ranging from a smiling face to a painful face. The child is told about the pain level of the faces on the scale and told to choose the face that best expresses his or her pain.

Child Fear Scale It was adapted from the Faces Anxiety Scale by McMurty and colleagues to measure fear in children undergoing painful medical procedures. The Child Fear Scale is a scale rated 0-4 that shows five hundred ranging from a neutral expression (0 = no worry) to a feared face (4 = serious anxiety).

Emotional Indicators Scale in Children: It is an easy-to-evaluate and easy-to-apply scale used to objectively define the emotional indicators that children show against medical procedures.

Collection of Data Two research-independent volunteer nurses with at least 10 years of experience will assist in the data collection process. The observer nurse will be informed by the researcher about the scale forms to be used in the study process. The polyclinic nurse will perform the routine nursing intervention. Nurses do not have conflicts of interest with research.

First of all, the participants who are waiting to have blood drawn at the entrance of the polyclinic by the researcher and who meet the sample selection criteria will be informed about the research and informed consent will be obtained from the child and parent. The data will then be recorded by asking questions about the characteristics of the participant and his/her parents included in the data collection form and the processing. Children who meet the criteria will be assigned to the application groups according to the randomization list created by the researcher.

Data evaluation/statistical methods of the study Descriptive statistics of the data; mean, standard deviation (median, minimum, maximum) will be given as frequency and percentage values. The assumption of normality of the quantitative data will be checked by the Shapiro-Wilk test. Unidirectional ANOVA (Bonferroni or Tukey test for binary comparisons) will be used for variables with normal distributions, while Kruskal-Wallis test (Dunn test for binary comparisons) will be used for variables that do not provide normality assumption. The correlation of quantitative data with each other will be evaluated by Pearson or Spearman's Rho correlation coefficients. The relationships between categorical variables will be examined by the Pearson Chi-square test or Fisher's Full probability test.

The data were analyzed using SPSS (22.0) software. The significance level was determined as 0.05 in all analyzes.

ELIGIBILITY:
Inclusion Criteria:

* Patient who needs to take intravenous blood
* The participant is in the 3-12 age group

Exclusion Criteria:

* Failure to obtain consent
* The child has an intellectual or neurological disability
* Failure to communicate in Turkish
* Having visual and hearing impairment
* The child has complaints such as pain, nausea, vomiting, etc. that disrupt his comfort due to another reason.
* 6 hours before the use of analgesic or sedative drugs
* Lack of healthy skin integrity
* Having repeated attempts
* Having syncope during blood collection

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
The Child Fear Scale | an average of 6 months
  Child Fear Scale (CSS) was used. This scale is a single-item self-report measure used to measure pain-related fear in children. This single-item scale consists of five gender-neutral facets. It ranges from a fearless (neutral) face on the far left to a face showing extreme fear on the far right. The evaluator's response indicates the level of fear. It can be used by parents and researchers before and during the procedure in children aged 5-10 years. CFS was applied to the children by the researcher to evaluate their fear levels regarding blood collection before, during and after the blood collection procedure.
Wong Baker Pain Scale | an average of 6 months
  Wong-Baker FACES (WB-FACES) Pain Rating Scale was used. This scale is used to rate pain intensity in children ages 3 and older. This numerical rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/no pain) to crying (10 = very painful). This scale was evaluated by the researcher during and after blood collection in this study.
Emotional Indicators Scale | an average of 6 months
  The Emotional Indicators Scale is used to assess the child's emotional reactions immediately after the needle enters the skin during blood collection. The scale measures emotional indicators such as crying, facial expressions, and distress, with ratings ranging from 0-5 (with 0 indicating no emotional response and 5 representing a strong emotional response). Higher scores on the scale may indicate a worse outcome in terms of emotional distress.This scale was evaluated by the researcher during blood collection in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Ülkü Güneş, Study Director — Faculty of Nursing Lecturer
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Kucuk Alemdar D, Yaman Aktas Y. The Use of the Buzzy, Jet Lidokaine, Bubble-blowing and Aromatherapy for Reducing Pediatric Pain, Stress and Fear Associated with Phlebotomy. J Pediatr Nurs. 2019 Mar-Apr;45:e64-e72. doi: 10.1016/j.pedn.2019.01.010. Epub 2019 Jan 30. PMID 30711327
- [Background] Arane K, Behboudi A, Goldman RD. Virtual reality for pain and anxiety management in children. Can Fam Physician. 2017 Dec;63(12):932-934. PMID 29237632
- [Background] Ballard A, Khadra C, Adler S, Doyon-Trottier E, Le May S. Efficacy of the Buzzy(R) device for pain management of children during needle-related procedures: a systematic review protocol. Syst Rev. 2018 May 22;7(1):78. doi: 10.1186/s13643-018-0738-1. PMID 29788987
- [Background] Binay S, Bilsin E, Gerceker GO, Kahraman A, Bal-Yilmaz H. Comparison of the Effectiveness of Two Different Methods of Decreasing Pain During Phlebotomy in Children: A Randomized Controlled Trial. J Perianesth Nurs. 2019 Aug;34(4):749-756. doi: 10.1016/j.jopan.2018.11.010. Epub 2019 Feb 20. PMID 30797673
- [Background] Burunsuz E.G, Köse S. (2020). The effect of butterfly patterned detection material used in intravenous catheter application on emotional and physiological indicators of children. Online Turkish Journal of Health Sciences, 5(4), (p:673-682).
- [Background] Çalış, H., Karataş, P. (2019). Atraumatic care approach in pediatric nursing: non-pharmacological applications in reducing pain, stress and anxiety. Koç University Journal of Education and Research in Nursing, 16 (3): (p:234-245). DOI:10.5222/HEAD.2019.234
- [Background] Çantaş Ayar, A. (2018). White noise during the process of taking blood from the heel of the foot in newborns, the effect of the position of the fetus in the lap and the fetal position given by hand on pain. Master's Thesis. Trabzon.
- [Background] Dalley JS, McMurtry CM. Teddy and I Get a Check-Up: A Pilot Educational Intervention Teaching Children Coping Strategies for Managing Procedure-Related Pain and Fear. Pain Res Manag. 2016;2016:4383967. doi: 10.1155/2016/4383967. Epub 2016 Apr 7. PMID 27445612
- [Background] Dincer, A. (2017). Fear: Language, Conceptualization, Cultural Dimension. International Journal of Turkish Literature Culture and Education, 6(2), (p:769-798).
- [Background] Dumandag, F. (2019). Evaluation of the effect of pre-procedure education on the compliance and anxiety level of the upper gastrointestinal tract endoscopy. Biruni University Institute of Health Sciences Department of Nursing Master's Program. Istanbul.
- [Background] Engin, M. (2020). A study to determine student opinions on the use of hologram technology in accounting education. Burdur Mehmet Akif Ersoy University, Institute of Social Sciences, Department of Accounting and Financial Management, Master's Thesis
- [Background] Gündüz, S., Yüksel, S., Aydeniz, G.E., Aydoğan, R.N., Türksoy, H., Dikme, İ.B., Efendiler, İ.(2016). Factors affecting the fear of hospitals in children. Journal of Child Health and Diseases, 59, (p:161-168).
- [Background] Khazar, D. (2021). Examination of the process of creating linear algebra concepts in three-dimensional hologram-assisted learning. Dokuz Eylül University, Institute of Educational Sciences, Department of Primary Education, PhD Thesis.
- [Background] Heden L, VON Essen L, Ljungman G. Randomized interventions for needle procedures in children with cancer. Eur J Cancer Care (Engl). 2009 Jul;18(4):358-63. doi: 10.1111/j.1365-2354.2008.00939.x. Epub 2008 Nov 27. PMID 19040458
- [Background] Heden L, von Essen L, Ljungman G. The relationship between fear and pain levels during needle procedures in children from the parents' perspective. Eur J Pain. 2016 Feb;20(2):223-30. doi: 10.1002/ejp.711. Epub 2015 Apr 2. PMID 25845466
- [Background] Helvaci, A. (2019). The role of artistic activities in overcoming children's fears of hospitals. Kocaeli University Journal of Fine Arts Faculty; 5(6), (pp. 24-30).
- [Background] Hologram technology? In which sector is it used? (2022, February 20). Access address:https://teknoloji.org/hologram-teknoloji-nedir-which-sektorlarda-kullaniyor/
- [Background] Inal, S., Canbulat, N. (2015). Use of Attention-Diverting Methods in Transactional Pain Management in Children. Current Journal of Pediatrics, 13(2), (p:116-121). Access address:https://doi.org/10.4274/jcp.29292
- [Background] İnci, R., Günay, U. (2019). Knowledge, Opinions and Applications of Pediatric Nurses for Therapeutic Play. Acıbadem University Journal of Health Sciences.10(3), (p:547-551. URL: https://doi.org/10.31067/0.2019.187
- [Background] Kayıkçı, Ş.,Yürekli, A. (2020). The use of hologram technology in video mobile communication. European Journal of Science and Technology, (p:94-99) . DOI: 10.31590/ejosat.779097
- [Background] Marashuna, O.(2011). Fears of medical procedures of secondary school students and influencing factors. Institute of Health Sciences, Near East University of the Turkish Republic of Northern Cyprus. Master's Thesis in Nursing. Cyprus.
- [Background] Ozel A, Cetin H. [Effects of vibrating tourniquet application on the pain felt for blood drawing in pediatric patients]. Agri. 2020 Jan;32(1):25-30. doi: 10.14744/agri.2019.04900. Turkish. PMID 32030695
- [Background] Pancekauskaite G, Jankauskaite L. Paediatric Pain Medicine: Pain Differences, Recognition and Coping Acute Procedural Pain in Paediatric Emergency Room. Medicina (Kaunas). 2018 Nov 27;54(6):94. doi: 10.3390/medicina54060094. PMID 30486427
- [Background] Sarman A, Sarman S, Tuncay S. (2021). Quantitative and content review of graduate theses made using virtual reality in nursing and published in YÖK Thesis. BUSAD; 2(2), (pp. 71 - 82).
- [Background] Semerci R, Kocaaslan EN, Akgun Kostak M, Akin N. [Reduction of pain during intravenous cannulation in children: Buzzy application]. Agri. 2020 Nov;32(4):177-185. doi: 10.14744/agri.2020.02223. Turkish. PMID 33398861
- [Background] Susam V, Friedel M, Basile P, Ferri P, Bonetti L. Efficacy of the Buzzy System for pain relief during venipuncture in children: a randomized controlled trial. Acta Biomed. 2018 Jul 18;89(6-S):6-16. doi: 10.23750/abm.v89i6-S.7378. PMID 30038198
- [Background] Sülü Uğurlu E.(2017). Nonpharmacological methods of pain relief in interventional procedures in children. Acıbadem University Journal of Health Sciences, 8(4),(p.198-201).
- [Background] Trost MJ, Chrysilla G, Gold JI, Mataric M. Socially-Assistive Robots Using Empathy to Reduce Pain and Distress during Peripheral IV Placement in Children. Pain Res Manag. 2020 Apr 9;2020:7935215. doi: 10.1155/2020/7935215. eCollection 2020. PMID 32351642
- [Background] Ye W, Zhang X, Li T, Luo C, Yang L. Mixed-reality hologram for diagnosis and surgical planning of double outlet of the right ventricle: a pilot study. Clin Radiol. 2021 Mar;76(3):237.e1-237.e7. doi: 10.1016/j.crad.2020.10.017. Epub 2020 Dec 9. PMID 33309030
- [Background] Yilmaz G, Alemdar DK. Using Buzzy, Shotblocker, and Bubble Blowing in a Pediatric Emergency Department to Reduce the Pain and Fear Caused by Intramuscular Injection: A Randomized Controlled Trial. J Emerg Nurs. 2019 Sep;45(5):502-511. doi: 10.1016/j.jen.2019.04.003. Epub 2019 Jun 27. PMID 31257044
- [Derived] Ozturk C, Gunes U. Reducing procedural pain and fear in children using a hologram fan and bubble machine: A randomized controlled trial of passive distraction techniques. J Pediatr Nurs. 2025 Dec 16;86:559-567. doi: 10.1016/j.pedn.2025.12.004. Online ahead of print. PMID 41406684
- See also: Wong-Baker Faces Pain Scale image, (2022, February 20) — https://www.ktu.edu.tr/dosyalar/farabikalite_86ee4.pdf
- See also: Hologram fan image, (2022, February 21st). — https://www.trendyol.com/hello/3d-hologram-fan-p-47404882